CLINICAL TRIAL: NCT00491231
Title: Is Orthostatic Hypotension Associated With Nondipping Hypertension
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Other Study IDs: SHEBA-07-4663-EG-CTIL
Record Dates: First submitted 2007-06-25; First posted 2007-06-26 (Estimated); Last update posted 2007-11-19 (Estimated); Status verified 2007-11

CONDITIONS: Orthostatic Hypotension; Nondipping Hypertension
Keywords: orthostatic hypotension; ambulatory blood pressure monitoring
MeSH Terms: conditions — Hypotension, Orthostatic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the study is to evaluate whether orthostatic hypotension is associated with nondipping hypertension.

Methods and patients: 400 subjects who are referred for 24hABPM will be filled questioner regarding their medical background and medications. All patients will be subjected to orthostatic test before connection to the 24 ABPM. The orthostatic changes in blood pressure and heart rate will be correlated to the changes in blood pressure and heart rate from day to night as recorded by the 24H ABPM.

ELIGIBILITY:
Inclusion Criteria:

* All patients who are referred for ABPM

Exclusion Criteria:

* Known secondary hypertension

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 400 subjects who are referred for 24hABPM
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2007-07; Study Completion 2008-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ehud Grossman, MD, Principal Investigator — The Chaim Sheba Medical Center
Locations (1):
- The Chaim Sheba Medical center, Tel Litwinsky, Ramat Gan, Israel